CLINICAL TRIAL: NCT03128203
Title: Effects of Intranasal Oxytocin on Striatal Functional Connectivity in Healthy Males
Brief Title: Effects of Intranasal Oxytocin on Striatal Functional Connectivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-36
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: Oxytocin; Resting-state; Functional connectivity; BOLD
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Oxytocin (Experimental)
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Oxytocin — Oxytocin, intranasally administrated
  Arms: Oxytocin
Drug: Placebos — Saline, intranasally administrated
  Arms: Placebo

SUMMARY:
To investigate whether 40 IU of intranasal oxytocin treatment can influence the resting-state functional connectivity in healthy males.

DETAILED DESCRIPTION:
In a double-blind, between-subject, placebo controlled design, investigators plan to investigate the effects of oxytocin treatment on resting-state functional connectivity.

Subject will receive either intranasal oxytocin or placebo administration and go through a seven-minute resting-state scan in MRI scanner to test whether oxytocin changes functional connectivity in the brain. Trait anxiety and mood questionnaires will be administered as control variables.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects without past or current psychiatric or neurological disorders

Exclusion Criteria:

* with MRI Contraindications

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 135 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Striatal functional connectivity alterations after drug administration | 45 minutes after drug administration
  fMRI-based resting state connectivity of the striatum will be compared between the oxytocin and the placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Becker, Dr., Principal Investigator — School of Life Science and Technology, University of Electronic Science and Technology of China
Locations (1):
- School of Life Science and Technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China